CLINICAL TRIAL: NCT01352910
Title: rTMS and Functional Paralysis
Acronym: PARALYSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/082/HP
Record Dates: First submitted 2011-05-11; First posted 2011-05-12 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Psychogenic Paralysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- effective rTMS (Experimental)
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator)
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — 120 pulses 0.2 Hz
  Arms: effective rTMS
Device: Sham rTMS — 120 pulses 0.2 Hz
  Arms: Sham rTMS

SUMMARY:
Psychogenic paralysis presents a real treatment challenge. Despite psychotherapy, physiotherapy, antidepressants, acupuncture or hypnosis, the outcome is not always satisfactory with persistent symptoms after long-term follow-up. In a preliminary retrospective study on 70 patients with psychogenic paralysis (44F/26M, mean age : 24.7 ± 16.6 ys), repetitive transcranial magnetic stimulation (rTMS) delivered over the motor cortex at low frequency was effective in 89% of cases (recovery: n=53, improvement: n=9), with an immediate or quasi-immediate recovery in 73% of patients (n=51).

We suggest that the dramatic improvement of psychogenic paralysis after rTMS could be due to the restoration of an appropriate cerebral connectivity by activating a suppressed motor cortex. Nevertheless, the possibility of a placebo effect cannot be ruled out.

A prospective multicentric (Rouen, Caen) randomized controlled trial versus placebo will be done for 94 patients with psychogenic paralysis, 1- to evaluate rTMS efficacy for paralysis at short and long term follow-up, and 2- to confirm rTMS safety. Two rTMS sessions will be performed at D0 and D1 (120 pulses over 2 days, delivered over the motor cortex at 2 Hz) with an active or a sham coil. Post-rTMS assessment will evaluate 1- the degree of the paralysis at D2 (quantified by a videotape) and D60 (quantified by an interview and a standardized examination), 2- the number and gravity of side effects.

If psychogenic paralysis improvement by motor cortex rTMS is confirmed, rTMS could be considered a useful early therapeutic option.

ELIGIBILITY:
Inclusion Criteria:

* Age > 14 years old
* Psychogenic paralysis according to the DSM-IV-R

Exclusion Criteria:

* Contra-indication of rTMS
* Pregnancy or breast-feeding
* Previous history of epilepsia
* Previous session of rTMS (for any indication)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Degree of paralysis at D2, quantified by a videotape made at D2 and interpreted by to independent examinators | D2

SECONDARY OUTCOMES:
Number of side effects occurred during the 2 days of rTMS, between D0 and D1 | D0, D1, D2
Degree of side effects gravity occurred during the 2 days of rTMS, between D0 and D1 | D0, D1 and D2
Degree of paralysis at D60, quantified by an interview and a standardized examination | D60

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Chastan, MD PhD, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Rouen University Hospital, Rouen